CLINICAL TRIAL: NCT04711954
Title: COVID-19 in People Living With HIV in Light of the 90-90-90 Goals: A Netherlands/Ukraine Research Collaboration.
Brief Title: HIV/COV in Ukraine-NL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Lviv Regional AIDS Health Center (Unknown)
Responsible Party: Principal Investigator, Casper Rokx, MD PhD, Erasmus Medical Center
Other Study IDs: 1990 Study
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Hiv; Covid19
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATHENA: Cohort of people living with HIV in the Netherlands
- LUKCY: Cohort of people living with HIV in the Lviv area, Ukraine

SUMMARY:
Contradicting preliminary results are available on the impact of COVID-19 in people with HIV (PWH). How achieving goals of the HIV 90-90-90 cascade of care influences the risk of COVID-19 in PWH is unclear. The primary objective is to determine the impact of COVID-19 in PWH cohorts from Ukraine and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

HIV infected No registered objection to use of data

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with HIV from patient cohorts in the Netherlands and Ukraine. All participants will be systematically included consecutively.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence COVID19 | Up to 2 years
  Prevalence (percent) of clinical COVID-19 in PWH cohorts from Ukraine and in the Netherlands.

SECONDARY OUTCOMES:
Incidence COVID-19 | Up to 2 years
  Incidence (nr cases/person years) of clinical COVID-19 cases in PWH cohorts from Ukraine and in the Netherlands
WHO categories COVID-19 | Up to 2 years
  Prevalence of no suspicion, possible, probable and proven COVID-19 cases in the past 6 months PWH cohorts from Ukraine and the Netherlands.
WHO categories COVID-19 | Up to 2 years
  Incidence of no suspicion, possible, probable and proven COVID-19 cases in the past 6 months PWH cohorts from Ukraine and the Netherlands.
WHO disease severity COVID-19 | Up to 2 years
  Proportion of COVID-19 patients according to the severity of COVID-19 on an adapted World Health Organisation 5 point disease severity scale (where 1=no symptoms, 2=symptoms but outpatient, 3=admitted to hospital, 4=admitted to ICU, 5=fatal) in people with HIV cohorts from Ukraine and the Netherlands.
Seroprevalence | Up to 2 years
  Anti-SARSCOV2 seroprevalence in PWH cohorts from Ukraine and the Netherlands
NPV/PPV WHO categories COVID19 | Up to 2 years
  Positive and negative predictive value of the WHO COVID-19 case probability categories on anti-SARSCOV2 serology in PWH cohort from Ukraine
Treatment | Up to 2 years
  Description of COVID-19 therapeutic management in PWH cohorts from Ukraine and the Netherlands
Predictors for COVID-19 | Up to 2 years
  Predictor variables for having clinical COVID-19 in PWH cohorts from Ukraine and the Netherlands according to 1) sex, 2) age categories (<50, 50-70, >70), 3) ART (LPV/r vs other and TDF containing vs non-TDF containing regimens), 4) most recent CD4+T-cell 5) HIV-RNA suppressed (<=50 / >50), 6) prior TB, 7) prior BCG, 8) HIV transmission group, 9) comorbidities (0 vs 1 vs >1).
Predictors for COVID-19 severity | Up to 2 years
  Predictor variables for the highest score on an ordinal scale for COVID-19 severity according to the adapted 5point WHO severity scale (where 1=no symptoms, 2=symptoms but outpatient, 3=admitted to hospital, 4=admitted to ICU, 5=fatal) in PWH cohorts from Ukraine and the Netherlands according to 1) sex, 2) age categories (<50, 50-70, >70), 3) ART (LPV/r vs other and TDF containing vs non-TDF containing regimens), 4) most recent CD4+T-cell 5) HIV-RNA suppressed (<=50 / >50), 6) prior TB, 7) prior BCG, 8) HIV transmission group, 9) comorbidities (0 vs 1 vs >1)

OTHER OUTCOMES:
HIV vs non-HIV | Up to 2 years
  Correlation of HIV status with the highest score on an ordinal scale for COVID-19 severity according to the adapted 5point WHO severity scale (where 1=no symptoms, 2=symptoms but outpatient, 3=admitted to hospital, 4=admitted to ICU, 5=fatal) in matched PWH cases with HIV uninfected controls by age, sex and comorbidities.
PPV/NPV WHO categories COVID-19 | Up to 2 years
  Positive and negative predictive value of the WHO COVID-19 case probability categories in the prior 3 months on anti-SARSCOV2 serology in PWH cohort from Ukraine
Effect of socio-economic status by questionnaire on COVID-19 incidence | Up to 2 years
  Evaluate the impact of social economic status on COVID-19 incidence.
Effect of socio-economic status on COVID-19 severity | Up to 2 years
  Evaluate the impact of social economic status on COVID-19 severity according to WHO 5 point scale (where 1=no symptoms, 2=symptoms but outpatient, 3=admitted to hospital, 4=admitted to ICU, 5=fatal)
Symptoms | Up to 2 years
  Describe symptoms associated with COVID probability in PWH cohorts from Ukraine and the Netherlands
Rapid Ag test | Up to 2 years
  Evaluate the PPV/NPV of the rapid antigen test in PWH with symptoms suspected of COVID-19 in Ukraine and the Netherlands

CONTACTS AND LOCATIONS:
Locations (2):
- Erasmus MC, Rotterdam, Netherlands
- Lviv Regional AIDS Health Center, Lviv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Other research group can contact the PI with a research question to gain access to IPD.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be kept up to 15 years

REFERENCES:
- [Derived] Vasylyev M, Buhiichyk V, Buhiichyck N, Groenendijk A, Ben I, Ostapiuk L, Sluzhynska M, Bierman WFW, van Kampen JJA, Wit FWNM, Reiss P, Rijnders BJA, Sluzhynska O, Rokx C. COVID-19 epidemiology and performance of the WHO clinical algorithm to diagnose COVID-19 in people with HIV from Ukraine. Int J STD AIDS. 2024 Jun;35(7):510-515. doi: 10.1177/09564624241231016. Epub 2024 Feb 6. PMID 38318789